CLINICAL TRIAL: NCT00271310
Title: The Effects of Long Term Inhalation of Hypertonic Saline in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Collaborators: Cystic Fibrosis Foundation (Other); National Health and Medical Research Council, Australia (Other); Cystic Fibrosis Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X95-0118B; 97/31391
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2006-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic

INTERVENTIONS:
Drug: hypertonic saline

SUMMARY:
The effect of long term inhalation of hypertonic saline in subjects with cystic fibrosis on lung function, incidence of respiratory tract infections, quality of life, quantitative microbiology and sputum cytokine profile. The hypothesis is that regular inhalation of nebulised hypertonic saline will have a beneficial effect on lung function and other clinical outcomes with no adverse effects on infection and inflammation in adults and children with cystic fibrosis.

DETAILED DESCRIPTION:
The study intervention is nebulised hypertonic (7%) saline (Active) or nebulised normal (0.9%) saline (Control) twice per day for 336 days. At a screening visit, subjects will complete quality of life questionnaires, be questioned regarding their medical history, undergo physical examination and spirometry, and will be requested to provide a sputum sample. The subject is then supervised taking their first dose to ensure the correct procedure is used and there are no adverse effects. The subject then commences taking the trial solution at home, and once a week completes a diary card to monitor factors such as respiratory tract infections and medication use. Subsequent visits are scheduled at Days 28, 84, 168, 252, 334, and 336, at which the same investigation are performed as at the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF (sweat tests/genotype)
* The subject, or their legal guardian for children under 18 years old, must provide written informed consent.
* The subject must be in stable clinical condition at the time of and for a period of 14 days prior to their recruitment into the study.
* Age > 6 years old
* FEV1 > 40% predicted for height, age and gender
* Proven or anticipated compliance with therapy or study protocol
* Regular attendee at a Cystic Fibrosis Clinic (> 2 visits per year)
* Able to reproducibly perform lung function tests (spirometry)
* Relatively stable nutritional status (< 2 kg weight loss in last 6 months and < 5 kg weight loss in last year)
* Known to have "normal" (for CF subject) laboratory tests - haematology, biochemistry, immunology, coagulation, etc.

Exclusion Criteria:

* Requiring home oxygen (pO2 <55mmHg or pCO2 >50mmHg) or assisted ventilation.
* Considered "terminally ill" or listed for transplantation (either lung or liver). Subjects that are listed for transplant after being enrolled in the trial are eligible to continue in the trial.
* Subjects colonised with Burkholderia cepacia. However, if a subject becomes colonised with B. cepacia during the trial, they should continue in the trial. Subjects should be considered to be B. cepacia positive if they have had even a single lifetime isolate. In these subjects, spirometry should be measured on a dedicated spirometer.
* Cigarette smoker.
* Exposure to investigational drugs within the past 30 days.
* Major haemoptysis (> 60 mL in a single episode) within the last twelve months.
* Concurrent illnesses eg. cor pulmonale, clinically significant liver disease (portal hypertension, varices).
* Known allergy to quinine sulphate, Glucose 6-phosphate dehydrogenase deficiency.
* Immune thrombocytopaenic purpura.
* Pregnant or lactating females.
* At risk females unwilling to use appropriate contraception to prevent pregnancy for the duration of their enrolment in the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164
Dates: Start 2000-09; Study Completion 2003-11

PRIMARY OUTCOMES:
Lung function (FEV1, FVC, FEF25-75)

SECONDARY OUTCOMES:
Pulmonary exacerbations (therapy-defined and symptom-defined)(number and duration)
Total antibiotic-days
Absenteeism
Weight / body mass index
Quality of life
Quantitative microbiology of sputum
Aquisition and loss of organisms from sputum
Cyotkine assays in sputum
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Peter T P Bye, PhD, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia

REFERENCES:
- [Result] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Derived] Wark P, McDonald VM, Smith S. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD001506. doi: 10.1002/14651858.CD001506.pub5. PMID 37319354